CLINICAL TRIAL: NCT00120107
Title: Tea's Effect on Atherosclerosis Pilot Study (TEA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kenneth Mukamal, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2003P000089; R21AT001899 (NIH)
Record Dates: First submitted 2005-07-07; First posted 2005-07-15 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Black Tea

SUMMARY:
The researchers propose a pilot study of the effect of long-term tea intake on atherosclerosis. Thirty patients at high risk for cardiovascular disease will be recruited and randomized to a six-month period of consumption of 3 cups per day of either tea, supplied as black tea solids readily dissolved in hot or cold liquid, or water.

At baseline and after 6 months, atherosclerosis in the aorta will be assessed using magnetic resonance imaging. The primary outcomes of this pilot study will be compliance with tea intake and 2 MRI examinations. As secondary outcomes, standard and novel cardiovascular risk markers, including inflammatory, prothrombotic, fibrinolytic, vascular and metabolic factors will be measured.

If successful, this pilot study will form the basis for a larger, long-term randomized trial to determine the effect of tea consumption on progression of atherosclerosis.

DETAILED DESCRIPTION:
Tea is widely thought to have health benefits, particularly on cardiovascular disease (CVD). The investigator's group recently found that intake of 2 or more cups of tea per day was associated with a 44% lower long-term mortality rate than abstention from tea among 1900 patients hospitalized with myocardial infarction. Short-term trials support a benefit of tea on endothelial function, but long-term randomized trials of tea intake on CVD and atherosclerosis are needed to test the effects of tea definitively.

The researchers propose a proof-of-principle pilot study of the effect of long-term tea intake on atherosclerosis. From a large hospital-based primary care practice, 30 patients at high risk for CVD will be recruited and randomized to a six-month period of consumption of 3 cups per day of either tea, supplied as black tea solids readily dissolved in hot or cold liquid, or water. The polyphenol content of these solids will be confirmed at baseline, and a single batch of tea throughout the study will be used. At baseline and after 6 months, aortic atherosclerosis using magnetic resonance imaging, an accurate and reproducible method for measurement of arterial plaque size, will be assessed. Adherence using urinary catechins, the primary flavonoids in tea, will be measured. The primary outcomes will be compliance with tea intake and 2 MRI examinations. As secondary outcomes, standard and novel cardiovascular risk markers, including inflammatory, prothrombotic, fibrinolytic, and metabolic factors will be measured. The researchers will also assess the effects of tea consumption on oxidizability of LDL and VLDL cholesterol, using a novel affinity-column chromatography approach, and on endothelial integrity, as assessed by serum markers of endothelial function. If successful, this pilot study will form the basis for a larger, long-term randomized trial to determine the effect of tea consumption on progression of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 55 years and the presence of either diabetes or two other cardiovascular risk factors. These risk factors will include hypertension, current smoking, LDL cholesterol ≥ 130 mg/dl, HDL cholesterol <40 mg/dl, or family history of premature coronary heart disease (as defined by Adult Treatment Panel III guidelines).

Exclusion Criteria:

* Patients with a history of congestive heart failure, myocardial infarction, arterial revascularization procedure (coronary, carotid, or peripheral), stroke, angina, or intermittent claudication will be excluded from this study. Either self-report or medical record evidence of these diagnoses will suffice for exclusion
* Intolerance or allergy to tea consumption
* Severe claustrophobia or intolerance to previous MRI examinations
* Standard MRI contraindications (for example, a pacemaker, intra-auricular implants, or intracranial clips)
* Severe illness expected to cause death or profound disability within six months
* Uncontrolled hypertension (blood pressure greater than or equal to 180/110)
* Chronic renal failure (serum creatinine >2.5 mg/dl or dialysis)
* History of hyponatremia in the last year (sodium <130 mEq/dl)
* Use of vitamin supplements greater than the recommended daily allowance
* Inability to speak English
* Lack of a working telephone

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-07; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The primary outcomes will be compliance with tea intake and 2 MRI examinations.

SECONDARY OUTCOMES:
Standard and novel cardiovascular risk markers, including inflammatory, prothrombotic, fibrinolytic, serum markers of endothelial function and metabolic factors. We will also assess oxidizability of LDL and VLDL cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Murray A Mittleman, MD, DrPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mukamal KJ, MacDermott K, Vinson JA, Oyama N, Manning WJ, Mittleman MA. A 6-month randomized pilot study of black tea and cardiovascular risk factors. Am Heart J. 2007 Oct;154(4):724.e1-6. doi: 10.1016/j.ahj.2007.07.008. PMID 17892999